CLINICAL TRIAL: NCT03528382
Title: The Impact of Early Cardiac Rehabilitation Quality Improvement System on the Incidence of Post-infarction HF: an Interventional Study
Brief Title: The Impact of Early Cardiac Rehabilitation of AMI Patients on the Incidence of Post-infarction HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu Bo (Other)
Responsible Party: Sponsor-Investigator, Yu Bo, Director, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016YFC1301105
Record Dates: First submitted 2018-05-07; First posted 2018-05-17 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- period I group (Experimental)
  Interventions: Behavioral: Cardiac rehabilitation quality improvement system
- period II group (Experimental)
  Interventions: Behavioral: Cardiac rehabilitation quality improvement system
- period III group (Experimental)
  Interventions: Behavioral: Cardiac rehabilitation quality improvement system

INTERVENTIONS:
Behavioral: Cardiac rehabilitation quality improvement system — Cardiac rehabilitation quality improvement system is divided into two period. The period I of rehabilitation has three parts, including daily life, rehabilitation exercise training, publicity and education. And the period II of rehabilitation is based on aerobic exercise, as well as combined with resistance and flexibility exercises

SUMMARY:
Background: Acute myocardial infarction (AMI) is the second cause of death worldwide. After AMI, the heart failure (HF) is a main cause of patient rehospitalization and death. Despite the total ischemic time of AMI is decreasing in general at present, the incidence of HF after AMI remains high. The incidence of HF in Switzerland and the United States are 25% and 14-16%, respectively, and the epidemiological statistic of AMI in the past 10 years was lacking in China, but the rate has been exceeded 22% by conservative estimation. Early cardiac rehabilitation quality improvement system has been shown to reduce incidence of post-infarction HF and improve cardiovascular function. However, early cardiac rehabilitation has low proportion and poor quality, which lacks of standard.

Objective: The purposes of this quality improvement study are to evaluate a pointed, two-phase intervention system to improve the proportion and quality of cardiac rehabilitation; to standardize the early cardiac rehabilitation procedure to improve the prognosis among patients with post-infarction HF.

Methods: Including the period I of cardiac rehabilitation, pre-discharge (baseline) assessment and the period II of cardiac rehabilitation.

Statistical analysis: Data analyses are performed using the software package SAS version 9.2 and all tests are 2-sided with P<0.05 denoting statistical significance. Quantitative data changes between groups which are compared with using the paired Student's t test and Wilcoxon rank sum test according to the data distribution, and categorical data is analyzed by chi-square test and ranked data is analyzed by Wilcoxon rank sum test. The investigator compare the incidence of heart failure in early rehabilitation patients between two phases according to the chi-square test of the rate of two groups, to explore the role of early cardiac rehabilitation after AMI in reducing the incidence of HF after AMI.

DETAILED DESCRIPTION:
Study design: After admission, and following clinical and diagnostic evaluation (12-lead electrocardiogram, Doppler echocardiography, symptom-limited cardiopulmonary exercise test and other related laboratory tests), all patients are discharged in low risk group (ejection fraction≥50% with AMI single-vessel lesion, emergency vascular recanalization without complication) and intermediate/high risk group (EF<50%, AMI partial blood transport reconstruction/multi-branch lesion, combined or uncombined with cardiogenic shock or heart failure). Researchers will assess inclusion and exclusion criteria, and patients who met the inclusion criteria need provide informed written consent in duplicate. All patients are enrolled in one I period rehabilitation during hospitalization and II period cardiac rehabilitation after discharge according to the different group. After 1 month, 2 months and 6 months, all patients undergo a telephone or outpatient follow-up assessment including training, smoking, drug usage and nutrient assessment. And after 3 months and 12 months, all patients undergo an outpatient follow-up assessment by 6-minute walking test and/or cardiopulmonary exercise test and three psychological scales (SF-12， GAD-7 and PHQ-9), besides the above.

The period I of cardiac rehabilitation: Patients who provide informed consents should assess indications and contraindications at first. The indications are: 1) no new emerging/repeated chest pain in 8 hours; 2) no further increase in the level of cardiac markers or cardiac enzymes (creatine kinase and troponin); 3) no obvious sign of decompensation of heart failure (the resting breath is difficult, combined with moist rale); 4) no new malignant arrhythmias or new electrocardiogram ischemic changes in the last 8 hours. The contraindications are: 1) hemodynamic instability or resting angina pectoris; 2) uncontrollable arrhythmia; 3) unable to rehabilitation due to disability or disease sequelae.

The period I of cardiac rehabilitation for low risk group is divided into five phases and each phase has three parts. The three parts are daily life (from complete rest in bed, low fat liquid diet to partly provided for themselves, low fat and semi-liquid diet to basically provided for themselves, low fat diet), rehabilitation exercise training (from passive joint exercises in bed to stand by bed and walk) and publicity and education (including introduction about cardiovascular intensive care unit, rehabilitation procedure, smoking cessation, risk factors of coronary heart disease, etc.). The period I of cardiac rehabilitation for intermediate/high risk group is divided into seven phases and each phase has three parts as well as the low risk group, but each part is more cautious than low-risk group.

Pre-discharge (baseline) assessment: One day before discharge, researchers should complete the assessment about patients who completed I period cardiac rehabilitation and fill in the cardiac rehabilitation quality feedback form. The assessments are as follows: 1) medical history assessment: recording patient medical history (coronary heart disease, hypertension, cerebrovascular disease, and/or peripheral vascular disease, hyperlipidemia, diabetes, congestive heart failure and chronic obstructive pulmonary disease, etc.); 2) physical examination: recording the heart rate, blood pressure and respiration of patients; checking whether there are engorgements of the neck veins, lung rale, cardiac souffle, arrhythmias and dropsy, etc; 3) accessory examination: recording the latest electrocardiogram and echocardiographic results); 4) nutrition assessment: assessing whether the patient is on high-fat diet or (and) high-salt diet and obese, setting a target weight based on BMI; 5) smoking assessment: assessing smoking status and let patients fill out the Fagerstrom test for nicotine dependence (FTND); 6) psychological assessment: let patients fill out the SF-12, GAD-7 and PHQ-9; 7) motor assessment: recording the maximum exercise load, the changes of heart rate and blood pressure from resting to maximum exercise load and rehabilitation process, terminal symptoms (angina and electrocardiogram abnormality), peak oxygen uptake, anaerobic threshold and alveolar air volume/carbon dioxide slope, through cardiopulmonary exercise test; 8) drug assessment: assessing and recording the name, dosage and usage of the drug; 9) adverse event assessment: assessing whether the patient with new or recurrent heart cerebral vascular disease, death and other adverse events when hospitalization, this part should be filled in the adverse event table; 10) Matters needing attention: Informing the patient or his family of precautions during the rehabilitation procedure and marking the doctor's contact number in the informed consent form, any hospitalization, reinfarction, or death should be immediately notified to the doctor.

The period II of cardiac rehabilitation: This period should last three months after discharge from the hospital. Exercise rehabilitation is based on aerobic exercise, and combined with resistance and flexibility exercises, including warm-up period (5-10 minutes), training period (20-40 minutes) and cool-down period (at least 5 minutes). Aerobic training should begin from discharge, at least 3 times per week and resistance training should begin in at least five weeks after AMI, 1 time per week at first. In addition, researchers should provide counseling about living habit and drug taking. Psychological counseling would be given to patients who have anxiety or depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 and ≤80 years old with a diagnosis of AMI (include ST segment elevated myocardial infarction and non-ST segment elevated myocardial infarction)

Exclusion Criteria:

* Pregnancy or lactation or with family planning during the trial;
* A history of heart failure;
* Severe liver dysfunction (The Alanine aminotransferase /aspartate aminotransferase level is over 3 times the upper normal limit);
* End-stage renal disease or creatinine plasma levels > 2.0mg/Dl;
* Tumor;
* AMI is caused by surgery, trauma, gastrointestinal bleeding or other complications caused by percutaneous coronary intervention;
* AMI occurred in patients who have been hospitalized for other reasons;
* Heart allograft transplantation;
* Participating in other clinical trials (except other subjects of this project) and have not reach the main end of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3103 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
The incidence of heart failure in 1 year follow-up | 1 year
  The incidence of heart failure after cardiac rehabilitate

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, MD,PhD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

REFERENCES:
- [Derived] Zheng X, Zhang M, Zheng Y, Zhang Y, Wang J, Zhang P, Yang X, Li S, Ding R, Siqin G, Hou X, Chen L, Zhang M, Sun Y, Wu J, Yu B. Quality indicators for cardiac rehabilitation after myocardial infarction in China: a consensus panel and practice test. BMJ Open. 2020 Dec 30;10(12):e039757. doi: 10.1136/bmjopen-2020-039757. PMID 33380480